CLINICAL TRIAL: NCT05012904
Title: Using Parental Involvement During Venipuncture to Reduce Venipuncture Pain and Anxiety in Children With Cancer: A Randomized Controlled Study
Brief Title: Using Parental Involvement During Venipuncture to Reduce Venipuncture Pain and Anxiety in Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Pınar BEKAR, Assistant Professor, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KAEK-792
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Anxiety; Cancer; Child; Nursing; Pain
MeSH Terms: conditions — Anxiety Disorders; Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: Randomization was done using the closed envelope method. A total of 60 cards with 30 "parent involvement" and 30 "control" labels were placed in sealed envelopes by the nurse who conducted the study. Children were asked to choose one of these envelopes and placed in the selected group. Children were randomized into two groups: a parent involvement group (n = 30) and a control group (n = 30).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent involvement Group (Experimental): A parent was involved in the procedure. The parent held the children in their arms and holding the extremity from which the blood was drawn, holding the hands of children and communicating with their children in the child's room, and in this way the parent was involved in the procedure.
  Interventions: Behavioral: parent involvement application
- Control Group (No Intervention): Routine venipuncture procedure was applied to the control group. The parent was present in the child's room but did not participate in the procedure.

INTERVENTIONS:
Behavioral: parent involvement application — A parent was involved in the procedure. The parent held the children in their arms and holding the extremity from which the blood was drawn, holding the hands of children and communicating with their children in the child's room, and in this way the parent was involved in the procedure.
  Arms: Parent involvement Group

SUMMARY:
This study aims to determine whether parental involvement during venipuncture reduces venipuncture pain and anxiety in children with cancer.

DETAILED DESCRIPTION:
This was a randomized controlled trial with parallel groups in which 60 children with cancer aged 6-12 were randomly allocated to a control group (n = 30) and a parent involvement group (n = 30). Each child's anxiety was evaluated by the child using the Children's Fear Scale before, during venipuncture, and each child's pain during the procedure was evaluated by the child using the Wong-Baker Faces Pain Rating Scale. Each child's heart rate and oxygen saturation were measured with a pulse oximeter device before, during the procedure.

Control group (n = 30): Routine venipuncture procedure was applied to the control group. The parent was present in the child's room but did not participate in the procedure.

Parent involvement group (n = 30): A parent was involved in the procedure. The parent held the children in their arms and holding the extremity from which the blood was drawn, holding the hands of children and communicating with their children in the child's room, and in this way the parent was involved in the procedure.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with cancer,
* requiring venipuncture for blood tests,
* 6-12 years old,
* not having taken any analgesics in the 6 hours before venipuncture,
* being in a non-terminal phase of the disease,
* absence of neutropenia,
* volunteering to participate in the study,
* the absence of any health problems that prevent communication in the parent or the child

Exclusion Criteria:

* reporting pain for another reason in the time of the venipuncture
* having another chronic disease besides cancer

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Wong-Baker FACES Pain Rating Scale (WB-FACES) | 3 MONTHS
  The Wong-Baker Faces Pain Rating Scale (WB-FACES) is used to evaluate pain levels in children. This numeric rating scale ranges from 0 to 10 and is represented by faces that display emotions ranging from smiling (0 = very happy or no pain) to crying (10 = the worst pain).

SECONDARY OUTCOMES:
Children's Fear Scale (CFS) | 3 MONTHS
  The Children's Fear Scale (CFS) is used to evaluate anxiety levels in children. It consists of five facial expressions representing a range from no anxiety (0) to severe anxiety (4).
Heart Rate | 3 MONTHS
  The heart rate and oxygen saturation values of the children in both groups were measured and recorded by the researcher before the procedure, during the procedure using a pulse oximeter device.
Oxygen Saturation | 3 MONTHS
  The heart rate and oxygen saturation values of the children in both groups were measured and recorded by the researcher before the procedure, during the procedure using a pulse oximeter device.

CONTACTS AND LOCATIONS:
Overall Officials: Emine EFE, Study Director — Akdeniz University, Department of Child Health and Disease Nursing
Locations (1):
- Pınar BEKAR, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No